CLINICAL TRIAL: NCT00877747
Title: Early Chemotherapy Intensification With BEACOPP in High-risk, Interim-PET Positive Advanced-stage Hodgkin Lymphoma:a GITIL Retrospective Multicenter Clinical Study
Brief Title: Early Chemotherapy Intensification in Interim-Positron Emission Tomography (PET) Positive Hodgkin Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ospedale Santa Croce-Carle Cuneo (Other)
Responsible Party: Principal Investigator, DR. ANDREA GALLAMINI, Professor, Ospedale Santa Croce-Carle Cuneo
Other Study IDs: HD-PET-intens-retr
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-10

CONDITIONS: Hodgkin Lymphoma
Keywords: PET
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PET2 negative: Patients with negative early interim PET after 2 courses of ABVD who continued therapy with ABVD
- PET2 positive: Patients with positive early interim PET after 2 courses of ABVD who changed their therapy to BEACOPP

SUMMARY:
Early interim-PET after two courses of chemotherapy is a powerful outcome predictor in advanced-stage Hodgkin Lymphoma (HL) patients treated with adriamycin (doxorubicin), bleomycin, vinblastine and dacarbazine (ABVD). Two-year Progression Free Survival of PET-2 positive patients is only 12%, but the optimal treatment for this patient subset is still unknown.

From January 2006 GITIL (Gruppo Italiano Terapie Innovative nei Linfomi) suggested an early intensification of chemotherapy with BEACOPP [Bleomycin, Etoposide, Adriamycin (doxorubicin), Cyclophosphamide, Oncovin (vincristine), Procarbazine, and Prednisone](4 escalated + 4 baseline cycles) for all the HL patients with a positive PET-2 after 2 ABVD courses. The investigators retrospectively recorded and analyzed these data in order to evaluate if this strategy could be of benefit for this subset of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced Hodgkin's lymphoma according to the World Health Organization classification
* Age 16-80
* Not previously treated
* Stage IIB to IVB or stage IIA with adverse prognostic factors (more than 3 nodal sites, ESR > 50 mm, bulky lesion)
* Written informed consent

Exclusion Criteria:

* Patients aged more than 80
* Concomitant or previously treated neoplastic disorder less than 5 years before the diagnosis of Hodgkin's lymphoma
* Psychiatric disorders
* Uncontrolled infectious disease
* Impaired cardiac (EF < 50%) or renal (creatinine clearance < 60 ml/m)function
* Pregnancy and lactation
* Uncompensated diabetes mellitus and fasting glucose levels over 200 mg/dl

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with advanced stage Hodgkin's lymphoma (IIB to IVB) or in stage IIA with adverse prognostic factors (more than 3 nodal sites, ESR > 50 mm, bulky lesion)
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2006-01; Primary Completion 2014-11 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years

SECONDARY OUTCOMES:
Incidence of progression/relapse | 2 years
Interim PET positive and negative predictive value | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gallamini, MD, Principal Investigator — Azienda Ospedaliera Santa Croce e Carle
Locations (1):
- Azienda Ospedaliera Santa Croce e Carle, Cuneo, Italy

REFERENCES:
- [Background] Gallamini A, Hutchings M, Rigacci L, Specht L, Merli F, Hansen M, Patti C, Loft A, Di Raimondo F, D'Amore F, Biggi A, Vitolo U, Stelitano C, Sancetta R, Trentin L, Luminari S, Iannitto E, Viviani S, Pierri I, Levis A. Early interim 2-[18F]fluoro-2-deoxy-D-glucose positron emission tomography is prognostically superior to international prognostic score in advanced-stage Hodgkin's lymphoma: a report from a joint Italian-Danish study. J Clin Oncol. 2007 Aug 20;25(24):3746-52. doi: 10.1200/JCO.2007.11.6525. Epub 2007 Jul 23. PMID 17646666
- [Derived] Gallamini A, Patti C, Viviani S, Rossi A, Fiore F, Di Raimondo F, Cantonetti M, Stelitano C, Feldman T, Gavarotti P, Sorasio R, Mule A, Leone M, Rambaldi A, Biggi A, Barrington S, Fallanca F, Ficola U, Chauvie S, Gianni AM; Gruppo Italiano Terapie Innovative nei Linfomi (GITIL). Early chemotherapy intensification with BEACOPP in advanced-stage Hodgkin lymphoma patients with a interim-PET positive after two ABVD courses. Br J Haematol. 2011 Mar;152(5):551-60. doi: 10.1111/j.1365-2141.2010.08485.x. Epub 2010 Dec 20. PMID 21166786